CLINICAL TRIAL: NCT00217828
Title: Effects of Citalopram on Hostility and CHD Risk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Treatment
Other Study IDs: 290; 2P01HL040962 (NIH)
Record Dates: First submitted 2005-09-19; First posted 2005-09-22 (Estimated); Last update posted 2014-06-11 (Estimated); Status verified 2014-06

CONDITIONS: Cardiovascular Diseases; Heart Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases | interventions — Citalopram

INTERVENTIONS:
Drug: citalopram

SUMMARY:
To evaluate the therapeutic effects of the serotonergic agent, citalopram, on hostility and other behavioral risk factors, and biological markers of disease risk (serum lipids, insulin and glucose; autonomic balance and stress-related cardiovascular reactivity; platelet activation).

DETAILED DESCRIPTION:
BACKGROUND:

Hostility, a broad personality dimension comprised of behavioral tendencies, cognitive biases and emotional or motivational characteristics appears to play an important role in the development of coronary heart disease (CHD). Furthermore, hostility apparently is important, not only as a function of its direct relationship to disease development, by virtue of its well documented link to a wide range of other risk factors, including life style factors (e.g., tobacco and alcohol use, imprudent diet), cardiovascular reactivity to stressful circumstances, and physiological indices (e.g., reactivity to acute stress, lipid levels, platelet activity, glucose regulation). It has been hypothesized that a common pathway underlying each of these factors is described by the serotonin system and by (dys) regulation of central serotonin pathways. Indeed, studies 1 and 2 of this program project application are devoted to an elaboration of this pathway as underlying behavioral, psychological, physiological and metabolic contributors to the development of CHD. The focus of this project is on the impact of short treatment with a selective serotonin reuptake inhibitor (SSRI) on hostility and the wide range of associated risk factors for CHD. Should this study prove successful, it will have the potential of significantly impacting treatment approaches that are aimed at reducing risk for the development and progression of CHD.

The study is one of four subprojects within a Program Project Grant entitled "Biobehavioral Studies of Cardiovascular Disease".

DESIGN NARRATIVE:

This is randomized placebo-controlled clinical trial of a select population, with the core questions revolving around the impact of brief (11 week) treatment with citalopram, a selective serotonin reuptake inhibitor (SSRI) on hostility as measured a number of ways. Healthy individuals who score above the median on standard measures of hostility will be identified. While questionnaire measures will be used to screen and select individuals, a host of measures of hostility will be employed to more fully capture the wide ranging aspects of this "personality" dimension, and thereby better ascertain the impact of the active agent. In addition to the measurement of the central personality dimension of interest, a wide range of other factors are to be measured. Life style risk factors measured include (e.g., the use of salivary cotinine to assess the validity of participants' self-report regarding tobacco use, the use of unannounced 24 hour dietary recalls, the use of pedometer to assess physical activity), autonomic activity (e.g., the wide range of indices available through the use of impedance cardiography, the use of heart rate variability, baroreceptor sensitivity), and platelet activity.

ELIGIBILITY:
No eligibility criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2002-03; Primary Completion 2003-02 (Actual); Study Completion 2003-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Kamarck (subproject PI) — University of Pittsburgh

REFERENCES:
- [Derived] Rice E, Vize C, Manuck S, Kamarck T. Mood reactivity to daily social conflict in hostile adults: An experimental intervention. Health Psychol. 2025 May;44(5):436-445. doi: 10.1037/hea0001411. PMID 40232779
- [Derived] Kamarck TW, Muldoon MF, Manuck SB, Haskett RF, Cheong J, Flory JD, Vella E. Citalopram improves metabolic risk factors among high hostile adults: results of a placebo-controlled intervention. Psychoneuroendocrinology. 2011 Aug;36(7):1070-9. doi: 10.1016/j.psyneuen.2011.01.005. Epub 2011 Feb 8. PMID 21306829